CLINICAL TRIAL: NCT05406258
Title: Self-Catheterization Mirror System for Female Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Megan O'Brien, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: STU00215439
Record Dates: First submitted 2022-06-01; First posted 2022-06-06 (Actual); Results first posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Self-Catheterization Mirror (Experimental): Following training, participants will have a modified mirror for self-catheterization. They will record the mirror used, position, and time for self-catheterization. They will also complete the System Usability Scale for each mirror related to self-operation and user satisfaction.
  Interventions: Device: Modified Self-Catheterization Mirror
- Standard Self-Catheterization Mirror (Active Comparator): Following training, participants will have a standard, hospital-provided mirror for self-catheterization. They will record the mirror used, position, and time for self-catheterization. They will also complete the System Usability Scale for each mirror related to self-operation and user satisfaction.
  Interventions: Device: Standard Self-Catheterization Mirror

INTERVENTIONS:
Device: Modified Self-Catheterization Mirror — Following training, participants will have a modified mirror for self-catheterization. They will record the mirror used, position, and time for self-catheterization. They will also complete the System Usability Scale for each mirror related to self-operation and user satisfaction.
  Arms: Modified Self-Catheterization Mirror
Device: Standard Self-Catheterization Mirror — Following training, participants will have a standard, hospital-provided mirror for self-catheterization. They will record the mirror used, position, and time for self-catheterization. They will also complete the System Usability Scale for each mirror related to self-operation and user satisfaction.
  Arms: Standard Self-Catheterization Mirror

SUMMARY:
The purpose of this study is to test a modified mirror system for female patients to use during self-catheterization.

DETAILED DESCRIPTION:
Many female patients have difficulties with self-catheterization. Mirrors currently used for this procedure have limited stability and visibility to easily view the urethral opening during catheterization, particularly for individuals with motor impairments. This can be especially frustrating because catheterization is performed frequently throughout the day and may need to occur at home or in public facilities.

The purpose of this study is to test the usability and efficacy of a modified self-catheterization mirror system for female patients. The modified self-catheterization mirror system makes adjustments to a standard, hospital-provided cathing mirror to help female patients with a range of motor abilities catheterize themselves in various postures and settings. Namely, the system offers (1) an alternative way to hold the mirror, by suspending it between the legs rather than attaching it to the toilet, and (2) lights that can be turned on for improved visibility during the self-catheterization process.

ELIGIBILITY:
Inclusion Criteria:

* Females age 13 or older
* Urinary retention related to spinal cord injury or other medical conditions resulting in need for catheterization
* Individuals with sufficient upper limb function to catheterize independently or with minimal assistance, or as deemed appropriate for the study by the Principle Investigator.

Exclusion Criteria:

* Individuals younger than 13 years old
* Individuals with cognitive deficits or visual impairments that may impact safe use of the devices used
* Severe Range of Motion restrictions of the upper and/or lower extremities
* Pregnant

Min Age: 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only one participant completed both arms of the study.
Period: Overall Study
Arm/Group | Modified Self-Catheterization Mirror | Standard Self-Catheterization Mirror
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Modified Self-Catheterization Mirror | Standard Self-Catheterization Mirror | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Customized [Count of Participants; unit: Participants] | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: System Usability Scale
Description: Patient-reported usability and experience when using the mirror, with scores ranging from -20 to +20 (higher scores indicating higher usability performance).
  This assessment included 10 items with statements that participants scored on a Likert scale from strongly disagree (-2) to strongly agree (+2).
Time Frame: This assessment was only completed once at the end of each arm within 3 days prior to inpatient discharge.
Measure: Number; unit: score on a Likert scale
Arm/Group | Modified Self-Catheterization Mirror | Standard Self-Catheterization Mirror
Number analyzed (Participants) | 1 | 1
score on a Likert scale | 4 | 7

2. Secondary Outcome: Time to Self-Cath
Description: Participants timed themself each time they used the during the study period. The time needed to set up the mirror and self-catheterize was averaged for all attempts during the study period.
Time Frame: 1-7 days
Measure: Mean (Full Range); unit: minutes
Arm/Group | Modified Self-Catheterization Mirror | Standard Self-Catheterization Mirror
Number analyzed (Participants) | 1 | 1
minutes | 13.81 [7 to 20] | 20 [20 to 20]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during active participation in the study (1-7 days).
Arm/Group | Modified Self-Catheterization Mirror | Standard Self-Catheterization Mirror
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-11-22): https://cdn.clinicaltrials.gov/large-docs/58/NCT05406258/Prot_000.pdf
  • Informed Consent Form (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/58/NCT05406258/ICF_001.pdf